CLINICAL TRIAL: NCT05521867
Title: Randomized Controlled Trial Comparing Endoscopic Balloon Dilation Versus Endoscopic Stricturotomy for Short Strictures (< 3 cm) Related to Crohn's Disease (the BEST-CD Trial)
Brief Title: Endoscopic Balloon Dilation Versus Endoscopic Stricturotomy for Short Crohn's Strictures
Acronym: BEST-CD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIG/IEC-BH&R 32 / 07.2022-05
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease
Keywords: Endoscopic balloon dilation; Endoscopic stricturotomy; Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic balloon dilation (Active Comparator): Confirmed Crohn's disease with gastro-duodenal or ileo-colonic short (<3 cm) strictures (both de novo and anastomotic) without prior history of endoscopic stricture therapy
  Interventions: Device: Endoscopic balloon dilation
- Endoscopic stricturotomy with or without stricturoplasty (Active Comparator): Confirmed Crohn's disease with gastro-duodenal or ileo-colonic short (<3 cm) strictures (both de novo and anastomotic) without prior history of endoscopic stricture therapy
  Interventions: Device: Endoscopic stricturotomy with or without stricturoplasty

INTERVENTIONS:
Device: Endoscopic balloon dilation — EBD procedures will be performed with wire guided CRE pneumatic balloon (controlled radial expansion balloon, Boston scientific, Marlborough, MA, USA 0of various sizes based on tightness of the stricture (10-12 mm, 12-15 mm, 15-18 mm, 18-20 mm) with graded dilations with inflation pressures varying from 3-8 ATM pressure. Balloon was inflated for at least 2 minutes and slowly deflated. A maximum of two sessions of dilation will be allowed with a minimum interval of 15-30 days between them.
  Arms: Endoscopic balloon dilation
Device: Endoscopic stricturotomy with or without stricturoplasty — Endoscopic stricturotomy would be done using either a triple-lumen needle-knife (Boston Scientific, Marlborough, MA) or with a electrosurgical IT knife2 (Olympus Medical Systems, Tokyo, Japan) in the setting of endoscopic retrograde cholangiopancreatography (ERCP) Endocut on Erbe medical device (USA Incorporated Surgical Systems, Marietta, GA) with the following electrocautery settings : Endocut Q (effect 3, cut duration 1, cut interval 3). Strictures will be incised in a circumferential or radial fashion until an adequate passage of the scope. Endoclips may be applied post stricturotomy to act as keep treated stricture open and to prevent delayed bleeding (referred as stricturoplasty). Choice of endoclips and decision to perform stricturoplasty would be at the discretion of endoscopist.
  Arms: Endoscopic stricturotomy with or without stricturoplasty

SUMMARY:
Crohn's disease (CD) related strictures can be treated endoscopically by endoscopic balloon dilation (EBD) or endoscopic stricturotomy (EST). EBD is is the established endoscopic treatment for short strictures in Crohn's disease. However, roughly half had recurrent symptoms and two third require surgery after EBD. ES have been used initially for endoscopic treatment of patients for whom EBD was unsuccessful. Subsequently it was shown that ES is a better modality for treating CD related strictures (specially short and anastomotic strictures) than EBD lowering the risk of future surgery and procedure related perforation albeit with an increased risk of bleeding. ES was shown to be non-inferior to re-do surgery in chronic pouch anastomotic sinus in ulcerative colitis (UC) and ileocolic anastomotic strictures in CD thus reducing surgical morbidity. However, these two modalities have not been compared in a randomized controlled manner. We aimed to compare the two endoscopic treatments with regard to clinical success, need for surgery or additional endoscopic procedure and safety in patients with CD who have short (<3 cm), predominantly fibrotic stenosis excluding those in the small bowel not accessible by endoscope/colonoscope.

DETAILED DESCRIPTION:
Study design: Single centre, open-label, randomised trial to be done in Asian Institute of Gastroenterology, India Study population: All eligible consecutive patients with CD who developed de-novo or anastomotic strictures will be included.

Study settings:

The proposed study would be conducted in a high volume tertiary GI centre (Asian Institute of Gastroenterology) performing nearly more than 200 endoscopic balloon dilation :EBD/Endoscopic stricturotomy: ES procedures per year with an well established inflammatory bowel disease (IBD) registry with more than 7000 IBD patients under follow up.

The study will be conducted after approval by the institutional ethics committee. Written informed consent would be taken from each participants and the study would conform to the 1975 Declaration of Helsinki ethical guidelines.

Data collection: A survey administration software (google forms) would be used to collect the participant data (age, sex, ethnicity, clinical features, smoking status, details of CD diagnosis, disease phenotype, extra intestinal manifestations, family history, history of intestinal resection, details of stricture diagnosis, details of stricture: degree, number, location, radiological finding: concurrent abscess, fistula, enhancement; drug history for CD, procedural details: technical success, symptomatic improvement, endoscopic improvement, stricture related emergency visit or hospitalization, complications, subsequent need for additional endoscopic procedures or surgery upto a follow up of 1 year). Follow-up details would be collected via physical visit or telephonic communication.

Technique and instruments: Endoscopic balloon dilation (EBD) procedures will be performed with wire guided controlled radial expansion (CRE) pneumatic balloon (controlled radial expansion balloon, Boston scientific, Marlborough, MA, USA of various sizes based on tightness of the stricture (10-12 mm, 12-15 mm, 15-18 mm, 18-20 mm) with graded dilations with inflation pressures varying from 3-8 atmosphere (ATM) pressure. Balloon was inflated for at least 2 minutes and slowly deflated. For mild ooze post EBD, balloon tamponade will also done with the same balloon. A maximum of two sessions of dilation will be allowed with a minimum interval of 15-30 days between them. Additional EBD sessions would be considered as additional endoscopic procedure for the purpose of the study.

Endoscopic stricturotomy would be done using a needle knife/insulted tip (IT) knife with the following electrocautery settings : Endocut Q (effect 3, cut duration 1, cut interval 3) as per by global interventional inflammatory bowel disease (IIBD) group consensus.

Definitions: Technical success for EBD was defined as ability to perform the EBD procedure. Scope passage after EBD/stricturotomy was assessed as a separate outcome which was defined as passage of endoscope through the area where EBD/ES was performed. This included colonoscope for colonic/pouch strictures, endoscope for upper GI and duodenal strictures and an enteroscope: motorized spiral or single balloon enteroscope for small bowel strictures except those in terminal ileum. Clinical success in EBD/ES was defined as clinical improvement in symptoms (pain/ intestinal, gastric outlet or colonic obstruction symptoms) after the procedure. Sustained clinical success was defined as absence of obstructive symptoms at 1 year follow up. Major adverse events were defined as perforation, bleeding requiring transfusion or any procedure related prolongation of hospitalization period or an endoscopic, radiologic or surgical intervention. Minor adverse events were bleeding not requiring blood transfusion, post procedural pain and any other self limiting complication (e.g., sore throat after spiral enteroscopy) which does not warrant prolongation of hospital stay. Adverse events will be recorded for all the patients; events were considered associated to be with the procedure when a causal association was possible, probable, or definite. Recurrence of symptoms would be defined as re-emergence of symptoms for which the procedure was initially performed.

Sample size Based on previous retrospective study, symptomatic improvement with EST and EBD (9.5% and 33.5% respectively, the estimated sample size is total 90 (45 in each group) keeping type 1 error as 0.05 and power as 80%.

Randomisation Patients will be randomly assigned (1:1) to receive either EBD (EBD group) or EST (EST group) using a digital en-block randomisation system (block size of four).

Data analysis Statistical analysis: Statistical analysis would be done by using statistical package for social sciences (SPSS, IBM: International Business machines, NY: New York, USA). Chi-square/Fisher's exact test was used to compare categorical variables and Mann-Whitney test would used to compare continuous variables between the two groups.P-value <0.05 would be considered statistically significant

Timeline: 3 years Recruitment of 100 CD patients with stenosis requiring EBD or EST over 2 years: follow up over 1 year.

Patient privacy An organised database for the purpose of this study will be formed based on google form with anonymised data set (i.e. name, address, and full post code will be removed, together with any other information which, in conjunction with other data held by or disclosed to the recipient, could identify the patient) which would be entered by clinical research assistant.

Study design Study type: Interventional (clinical trial) Estimated enrolment: 100 patients Allocation: Randomized Intervention model: Parallel assignment Masking: none (open label) Primary purpose: Therapeutic Official title: Randomized controlled trial comparing endoscopic balloon dilation versus endoscopic stricturotomy for short strictures (< 3 cm) related to Crohn's disease (the BEST-CD trial) Estimated start date : August - September 2022 (after ethical approval) Estimated recruitment completion: July - August 2023 Estimated study completion date: July - August 2023

ELIGIBILITY:
Inclusion criteria Primary confirmed diagnosis of CD with obstructive symptoms

1. Gastro-duodenal and ileo-colonic strictures (both de novo and anastomotic strictures)
2. Short strictures (<3 cm)
3. Fibrotic or mixed stricture (predominantly fibrotic)
4. Strictures treated with either EST or EBD.

Exclusion Criteria:

1. No established diagnosis of CD;
2. No endoscopic therapy; and
3. A combination therapy of EST and EBD at the onset
4. Small bowel CD related stricture requiring enteroscopy guided dilation
5. Predominantly ulcerated strictures (mixed or pure ulcerated strictures)
6. Long strictures (>3 cm)
7. Pediatric Patients (<18 years)
8. Pregnant or lactating mother
9. Not willing to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of the percentage of sustained clinical improvement in EBD and ES arms | 1 year
  To compare sustained clinical improvement post EBD and ES (%) (time frame :
  1year): percentage of patients having no obstructive symptoms due to CD related stenosis for which EBD/ES was performed for a period of 1 year

SECONDARY OUTCOMES:
Comparison of the percentage of patients requiring additional interventions in EBD and ES arms | 1 year
  To compare need for additional intervention (EBD/EST/Surgery) between EST and EBD arm (%) : the percentage of patients who require additional interventions for CD related stenosis over period of 1 year
Comparison of percentage of technical success in EBD and ES arms | During procedure
  To compare technical success between EBD and ES (%): Percentage of patients in whom endoscope is passable after EBD/ES
Comparison of the percentage of stricture related emergency department visits in EBD and ES arms | 1 year
  To compare stricture related visit to the emergency department after EST versus EBD: percentage of patients visiting the emergency department for CD stenosis related symptoms post EBD/ES over period of 1 year
Comparison of the percentage of patients requiring stricture related hospitalizations in EBD and ES arms | 1 year
  To compare structure related hospitalization with EST versus EBD: percentage of patients visiting undergoing hospitalization for CD stenosis related symptoms post EBD/ES over period of 1 year
Comparison of the percentage of procedure related complications related to EST versus EBD | 1 month
  To compare complications related to EST versus EBD as per American Society of Gastrointestinal Endoscopy (ASGE) lexicon for adverse seventh during endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Partha Pal, MD, DNB, Principal Investigator — Asian lnstitute of Gastroenterology
Locations (1):
- Asian lnstitute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-07-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT05521867/Prot_000.pdf
  • Informed Consent Form (2022-07-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT05521867/ICF_001.pdf